CLINICAL TRIAL: NCT05200182
Title: fNIRS-based Neurofeedback Intervention for Cognitive Control Improvement in Emotional Overeating
Acronym: Cemov
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 35RC20_9849_Cemov; 2021-A02314-37 (Other: ID-RCB)
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Hyperphagia
Keywords: emotional overeating; functional near infraRed spectroscopy; neurofeedback; cognitive control
MeSH Terms: conditions — Hyperphagia | interventions — Neurofeedback; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study A (Other): Validation of the reward system-related fMRI task, as determined by an increased activation on the brain reward structure (striatum) under the task.
  Interventions: Device: Neurofeedback with functional near infra-red spectroscopy; Device: resting-state fMRI; Device: Electro gastrogram
- Study B - Neurofeedback (Experimental): The neurofeedback protocol will be the same during the 8 sessions constituting the protocol and taking place over a period of 4 weeks (2 neurofeedback sessions per week, the first and the last one in an MRI context). It will last 15 minutes per session, and during each session, the volunteer will have to increase the brain activity of his/her dlPFC using a visual gauge representing the "activity level" of his/her own dlPFC. No specific instructions will be given to the volunteer so that he/she can develop his/her own internal strategy to increase this "activity level".
  Interventions: Device: Neurofeedback with functional near infra-red spectroscopy; Other: oral microbiota collection; Other: Questionnaires; Device: resting-state fMRI; Device: Electro gastrogram; Behavioral: Emotional Stroop task
- Study B - Control (Sham Comparator): In the control group with neurofeedback sham, the participants will receive the same instruction but will be shown a random signal, the goal being that the control strategy the participant tries to implement is not correlated with the visual feedback provided by the gauge.
  Interventions: Device: Sham Neurofeedback; Other: oral microbiota collection; Other: Questionnaires; Device: resting-state fMRI; Device: Electro gastrogram; Behavioral: Emotional Stroop task

INTERVENTIONS:
Device: Neurofeedback with functional near infra-red spectroscopy — the neurofeedback protocol will last 15 minutes per session, and during each session, the volunteer will have to increase the brain activity of his/her dorsolateral prefrontal cortex using a visual gauge representing the "activity level" of his/her own dorsolateral prefrontal cortex. No specific instructions will be given to the volunteer so that he/she can develop his/her own internal strategy to increase this "activity level".
  Arms: Study A; Study B - Neurofeedback
Device: Sham Neurofeedback — the participants will receive the same instruction but will be shown a random signal
  Arms: Study B - Control
Other: oral microbiota collection — an examination and oral swab for oral microbiota analysis will be performed by a dentist
  Arms: Study B - Control; Study B - Neurofeedback
Other: Questionnaires — questionnaires for pre-intervention behavioral characterization
  Arms: Study B - Control; Study B - Neurofeedback
Device: resting-state fMRI — characterize the brain function of volunteers by resting-state fMRI
Device: Electro gastrogram — Volunteers will also be equipped with an MRI-compatible electro-gastrogram device to correlate gastric signals with brain activity during rsMRI acquisition.
Behavioral: Emotional Stroop task — an emotional Stroop task adapted to food and body image representation
  Arms: Study B - Control; Study B - Neurofeedback

SUMMARY:
Emotional overeating is characterized by an excessive food intake in the context of intense emotional situations, such as acute stress one. Emotional overeating, as a behavioral trait, can increase the risk of to develop eating disorders or eating-related diseases, such as metabolic syndrome, obesity, type-2 diabetes. Recently, imaging modalities, such as magnetic resonance imaging (MRI) and electro-encephalography (EEG), have been adapted in order to perform neurofeedback consisting on presenting the brain activity instantaneously to the participant, that give him the possibility to modify this activity by his own mean. Neurofeedback has already shown some efficacy, either with explicit or implicit instruction.

Compared with functional MRI (fMRI), functional near infra-red spectroscopy (fNIRS) is easy to handle, less expensive, and does not require a lying position. fNIRS is consequently more adapted for repeated acquisitions. Neurofeedback has already shown some promising results for neurological and psychiatric diseases. For mental states and emotion regulation, neurofeedback targeting the prefrontal cortex (PFC) has also shown promising outcomes. In this project, the investigators want to assess the effect of neurofeedback targeting the dorsolateral PFC (dlPFC) in a population of young adult women presenting emotional overeating. The investigators aim to improve the cognitive control and to reduce the episodes of emotional overeating in order to prevent the occurrence of subsequent pathologies.

The intervention effect will be characterized with: (i) fMRI in order to evaluate the effect on cognitive control (with resting state fMRI or rsMRI) and on the reward system; (II) questionaries directly and one month after intervention in order to assess the behavioral effect.

Besides an expected effect on emotional overeating, the investigators will evaluate whether an improvement of cognitive control can also promote positive effect on other behavioral traits that could lead to some pathologies such as food addiction.

As a prerequisite to this study on emotional overeating (study B), the investigators will firstly validate on healthy subjects (study A) a reward anticipation fMRI task, which will be further used in study A in order to characterized the effect of neurofeedback on the reward system.

ELIGIBILITY:
Eligibility

Study A :

* Minimum age : 18 Years
* Maximum Age : 50 Years
* Sex : women or men

Inclusion Criteria :

* Normal Body Mass Index (18.5-25),
* Right-handlers
* Affiliated to a social security scheme
* Having given a free, informed and written consent

Exclusion Criteria :

Related to the study - Insufficient command of French

Related to Magnetic Resonance Imagine

* Implantable cardiac pacemaker or defibrillator;
* Neurosurgical clips;
* Cochlear implants;
* Neural or peripheral stimulator;
* Foreign orbital or brain metallic foreign bodies;
* Endoprostheses implanted for less than 4 weeks and osteosynthesis materials placed for less than 6 weeks;
* Claustrophobia. Related to near infra Red spectroscopy
* Hairs that do not allow proper near infra Red spectroscopy measurement upon ligh blockage

Study B

* Minimum age : 18 Years
* Maximum Age : 25 Years
* Sex : women

Inclusion Criteria :

* Normal BMI (18.5-25),
* Right-handlers
* Affiliated to a social security scheme
* Having given a free, informed and written consent
* Based on emotional overeating questionary : having emotional overeating episodes > 6 days in a month for at least one negative emotion

Exclusion Criteria :

Related to the study

* Insufficient command of French
* Excessive consumption of alcohol or other psychoactive substances (determined on the basis of the Alcohol Use Disorders Identification Test questionnaires - excluded if score > 12 and "Car, Relax, Alone, Forget, Friends, Trouble" questionnaire - excluded if score> 1 " yes ")
* Eating disorders ("sick, control, one stone, fat, food" questionnaire >2)
* Food addiction (Yale Food Addiction Score 2.0, score >2
* With psychoactive treatment
* Digestive or gastric disorders

Related to magnetic resonance imaging

* Implantable cardiac pacemaker or defibrillator;
* Neurosurgical clips;
* Cochlear implants;
* Neural or peripheral stimulator;
* Foreign orbital or brain metallic foreign bodies;
* Endoprostheses implanted for less than 4 weeks and osteosynthesis materials placed for less than 6 weeks;
* Claustrophobia.

Related to near infraRed spectroscopy

- Hairs that do not allow proper near infraRed spectroscopy measurement upon ligh blockage

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change in cortico-striatal connectivity | 4 weeks
  Significant change in cortico-striatal connectivity as determined with resting state functional magnetic resonance imaging correlation coefficient between the first magnetic resonance imaging and the last magnetic resonance imaging visit

CONTACTS AND LOCATIONS:
Overall Officials: Romain Moirand, MD, Principal Investigator — CHU Rennes
Locations (1):
- Chu Rennes - Pontchaillou, Rennes, France